CLINICAL TRIAL: NCT05341817
Title: The Use of Letrozole or Mifepristone for Pretreatment of Medical Termination of Pregnancy: a Randomized, Non-inferiority Trial
Brief Title: The Use of Letrozole or Mifepristone for Pretreatment of Medical Termination of Pregnancy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Seet Meei Jiun, Assistant Professor, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB 202110-00035
Record Dates: First submitted 2022-04-05; First posted 2022-04-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Abortion in First Trimester
Keywords: Medical termination of pregnancy; Abortion; Induced; mTOP; letrozole; mifepristone; misoprostol
MeSH Terms: interventions — Letrozole; Mifepristone

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The treatment doctor during the Day 21-28 follow-up visit will be blinded to the treatment allocation of the study participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole (Experimental): Day 1: Oral letrozole 10mg under direct observation therapy (DOT) in the clinic Day 2: Oral letrozole 10mg to self-administer at home Day 3: Oral letrozole 10mg to self-administer at home or at the hospital. Vaginal misoprostol 800mcg given in the ward, followed by vaginal misoprostol 400mcg, approximately 4 hours later, if subject showed no signs of abortion
  Interventions: Drug: Letrozole
- Control (Active Comparator): Day 1: Oral mifepristone 200mg (control) under direct observation therapy (DOT) in clinic Day 2: NIL medication to be self-administered at home Day 3: NIL medication to be self-administered at home. Vaginal misoprostol 800mcg given in the ward, followed by vaginal misoprostol 400mcg, approximately 4 hours later, if subject showed no signs of abortion
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Letrozole — Letrozole priming before mTOP is used as an alternative to the use of mifepristone. Women randomly assigned (1:1) to the Letrozole arm will receive 10 mg letrozole daily for 3 days followed by 800 μg misoprostol.
  Arms: Letrozole
Drug: Mifepristone — Mifepristone priming before mTOP is the current standard of care. Women randomly assigned (1:1) to the Control arm will receive 200 mg mifepristone followed by 800 μg misoprostol 2 days later.
  Arms: Control

SUMMARY:
Medical termination of pregnancy (mTOP) generally involves using either a combined regimen consisting of mifepristone and misoprostol, or a misoprostol-only regimen. Complete abortion rates of first trimester mTOP with the use of misoprostol-only regimen varies between 74-88%. With the addition of mifepristone as pre-treatment drug, this improves success rates to 93-97%. Mifepristone, an anti-progesterone, is relatively expensive and is subject to stringent regulations for usage in addition to restricted access in many countries. Therefore, there is a need to find a cheaper and more readily available, yet effective alternative.

The use of letrozole (an aromatase inhibitor) in mTOP is postulated to suppress estradiol levels (an important factor in the maintenance of early pregnancy), therefore enhancing the effect of misoprostol in inducing abortion. Studies have shown that pre-treatment with letrozole achieves a complete abortion rate of 77-98%, similar to that in mifepristone-Misoprostol studies.

The investigators hypothesise that letrozole is equivalent to mifepristone for the pre-treatment of mTOP and propose to conduct a randomised, non-inferiority trial for mTOP up to 10 weeks gestation with two arms as detailed below:

1. Oral letrozole 10mg daily for 3 days, followed by vaginal misoprostol on Day 3 (Intervention group)
2. Oral mifepristone 200mg once on Day 1, followed by vaginal misoprostol 800mcg on Day 3. Then, 4 hours later, another dose of 400mcg PV misoprostol if no signs of abortion (Control group - current practice).

The investigators aim to include a total of 144 patients, 72 in each arm, to detect a non-inferiority margin of 15% with a power of 80% at 5% significance. The investigators primary outcome will be rate of complete abortion by Day 21-28 of mTOP.

This pilot RCT will provide preliminary data and preparation for larger grant application which will provide necessary evidence to enhance the care of women undergoing mTOP, with enhanced cost-savings and availability.

DETAILED DESCRIPTION:
The standard of care for termination of pregnancy (TOP) has shifted from a predominantly surgical approach towards medical strategy. Medical termination of pregnancy (mTOP) has increased in popularity worldwide as it is cost savings, non-invasive and there is avoidance of risks associated with surgery.

In general, mTOP involves using either a combined regimen consisting of mifepristone and misoprostol which is the current gold standard of care, or a misoprostol-only regimen. The World Health Organisation (WHO) recommends the use of mifepristone for pre-misoprostol priming when mifepristone is available, and the alternative of misoprostol-only when mifepristone is not accessible. Compared with misoprostol alone, pre-treatment with mifepristone followed by misoprostol has been shown to improve the success rate of complete abortion. However, the widespread use of mifepristone is limited by the high cost of therapy and unavailability in many countries. Hence, there is an urgent unmet need for a cheaper and more readily available alternative.

Letrozole priming before mTOP has been proposed as an alternative to the use of mifepristone. The proposed mechanism is a reduction in serum estrogen levels, leading to a concomitant reduction in progesterone receptor concentration necessary for the maintenance of pregnancy. Several randomised controlled trials (RCTs) have been performed by comparing the effectiveness of using letrozole for mTOP priming before misoprostol versus misoprostol alone. The combination of letrozole with misoprostol has shown to be effective in improving the success rates of complete abortion up to 10 weeks gestation, compared with misoprostol alone. Given its low price, ready availability worldwide and common usage in the fields of ovulation induction and breast cancer, letrozole may be a potential alternative to mifepristone in mTOP priming. While medication costs vary from country to country, the cost of a course of letrozole is largely cheaper than mifepristone. Unfortunately, no study has been designed to specifically compare the effectiveness of letrozole versus mifepristone pre-treatment regimes in the management of mTOP. Independent examination of the pre-treatment effects of letrozole and misoprostol versus misoprostol alone in different studies (different population characteristics) restricted valid comparison between treatments. This forms the key motivation for the investigators' proposed study.

To address the aforementioned knowledge gaps, this study aims to conduct a non-inferior RCT to investigate whether pre-treatment with letrozole before misoprostol is comparable to mifepristone pre-treatment before misoprostol mTOP in patients up to 10 weeks gestation. Women will be randomly assigned (1:1) to either receive 10 mg letrozole daily for 3 days followed by 800 μg misoprostol, or 200 mg mifepristone followed by 800 μg misoprostol 2 days later. This RCT is designed as a non-inferiority trial. Thus, the investigators expect that no significant differences in abortion outcomes will be observed between the two groups.

The primary outcome is complete abortion rates. Secondary outcomes include time-to-abortion interval, the number of misoprostol doses required, healthcare resource utilisation and side effects.

Specific Aim 1: To compare complete abortion rates at day 21-28 of mTOP in patients using letrozole/misoprostol regime versus mifepristone/misoprostol regime. The investigators hypothesise that letrozole will achieve similar complete abortion rates as mifepristone when used as priming of mTOP. Complete abortion will be defined as no further intervention required e.g. medical or surgical treatment for retained products of conception.

Specific Aim 2: To determine if letrozole/misoprostol regime results in better healthcare resource utilisation than mifepristone/misoprostol regime. The investigators hypothesise that letrozole is a resource-efficient alternative as measured by length of hospital stay, need for emergency department attendance and need for additional medical/surgical treatment.

The successful completion of this RCT will provide the data necessary to show the non-inferiority of letrozole compared against mifepristone. This will lead to the introduction of a more cost-effective and more accessible mTOP service for patients, as letrozole is cheaper and more widely available as compared to mifepristone. The expansion of mTOP regimes may help to save hospital resources with less reliance on surgical methods (manpower and expertise, logistics, and cost etc.) in the long run.

ELIGIBILITY:
Inclusion Criteria:

* 21 years and above
* Patient requesting for medical termination of pregnancy (mTOP)
* Patient eligible for legal abortion according to the Termination of Pregnancy Act (Chapter 324)
* Gestational age ≤10 weeks (on day 1 of mifepristone or letrozole administration) as confirmed by the first trimester dating scan
* Singleton pregnancy
* Patient is agreeable to undergo surgical evacuation or repeat medical therapy if treatment fails
* Willing and able to provide written, informed consent

Exclusion Criteria:

* History or evidence of adrenal pathology, steroid-dependent cancer, porphyria, poorly controlled hypertension, bronchial asthma, thromboembolism and severe cardiac/renal/liver disease
* Haemoglobin level of <9.5 g/L
* Presence of an intrauterine contraceptive device
* Breastfeeding
* Reported allergic reaction to mifepristone, misoprostol or letrozole,
* Participating in another trial of investigational medicinal products during the current pregnancy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of complete abortion by Day 21-28 | Day 21-28 of study procedure
  Rate of complete abortion by Day 21-28 (defined as no further intervention required e.g. medical or surgical treatment for retained products of conception)

SECONDARY OUTCOMES:
Number of patients who require surgical evacuation of uterus for retained product of conception (POC) | Day 1-28 of study procedure
Number of patients who require repeated medical therapy for retained product of conception (POC) | Day 1-28 of study procedure, After Day 28 of study procedure
Number of doses of misoprostol administered for expulsion of product of conception (POC) | Day 3-4 of study procedure
Time interval between administration of first dose of misoprostol and expulsion of product of conception (POC) | Day 3-4 of study procedure
Number of patients who need blood transfusion | Day 1-28 of study procedure, After Day 28 of study procedure
Number of patients who require analgesia according to the analgesic ladder | Day 1-4 of study procedure
Number of patients who experience minor side effects including pain, bleeding, fever, vomiting and diarrhoea | Day 1-28 of study procedure, After Day 28 of study procedure
Length of hospital stay | Day 1-28 of study procedure, After Day 28 of study procedure
Number of patients who require unscheduled emergency department visit or hospital admission | Day 1-28 of study procedure, After Day 28 of study procedure
Number of patients who develop severe allergic reactions | Day 1-28 of study procedure, After Day 28 of study procedure
Number of adverse events reported | Day 1-28 of study procedure, After Day 28 of study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Meei Jiun Seet, Principal Investigator — Consultant at KK Women's and Children's Hospital, Singapore
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedgh G, Bearak J, Singh S, Bankole A, Popinchalk A, Ganatra B, Rossier C, Gerdts C, Tuncalp O, Johnson BR Jr, Johnston HB, Alkema L. Abortion incidence between 1990 and 2014: global, regional, and subregional levels and trends. Lancet. 2016 Jul 16;388(10041):258-67. doi: 10.1016/S0140-6736(16)30380-4. Epub 2016 May 11. PMID 27179755
- [Background] Medical management of abortion. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK536779/ PMID 30702834
- [Background] Abubeker FA, Lavelanet A, Rodriguez MI, Kim C. Medical termination for pregnancy in early first trimester (</= 63 days) using combination of mifepristone and misoprostol or misoprostol alone: a systematic review. BMC Womens Health. 2020 Jul 7;20(1):142. doi: 10.1186/s12905-020-01003-8. PMID 32635921
- [Background] Creinin MD, Shore E, Balasubramanian S, Harwood B. The true cost differential between mifepristone and misoprostol and misoprostol-alone regimens for medical abortion. Contraception. 2005 Jan;71(1):26-30. doi: 10.1016/j.contraception.2004.07.011. PMID 15639068
- [Background] Shi L, Shi SQ, Given RL, von Hertzen H, Garfield RE. Synergistic effects of antiprogestins and iNOS or aromatase inhibitors on establishment and maintenance of pregnancy. Steroids. 2003 Nov;68(10-13):1077-84. doi: 10.1016/j.steroids.2003.09.002. PMID 14668001
- [Background] Lee VC, Gao J, Lee KF, Ng EH, Yeung WS, Ho PC. The effect of letrozole with misoprostol for medical termination of pregnancy on the expression of steroid receptors in the placenta. Hum Reprod. 2013 Nov;28(11):2912-9. doi: 10.1093/humrep/det345. Epub 2013 Aug 26. PMID 23980056
- [Background] Lee VC, Yeung TW, Tang OS, Ng EH, Yeung WS, Ho PC. Effect of letrozole on uterine artery Doppler flow indices prior to first-trimester termination of pregnancy: a randomized controlled trial. Ultrasound Obstet Gynecol. 2012 Oct;40(4):392-7. doi: 10.1002/uog.11115. PMID 22302719
- [Background] Yung SSF, Lee VCY, Chiu PCN, Li HWR, Ng EHY, Yeung WSB, Ho PC. The effect of 7 days of letrozole pretreatment combined with misoprostol on the expression of progesterone receptor and apoptotic factors of placental and decidual tissues from first-trimester abortion: a randomized controlled trial. Contraception. 2016 Apr;93(4):323-330. doi: 10.1016/j.contraception.2015.12.005. Epub 2015 Dec 19. PMID 26707996
- [Background] Lee VCY, Ng EHY, Yeung WSB, Ho PC. Misoprostol with or without letrozole pretreatment for termination of pregnancy: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):317-323. doi: 10.1097/AOG.0b013e3182073fbf. PMID 21252745
- [Background] Nash CM, Philp L, Shah P, Murphy KE. Letrozole pretreatment prior to medical termination of pregnancy: a systematic review. Contraception. 2018 Jun;97(6):504-509. doi: 10.1016/j.contraception.2017.11.003. Epub 2017 Nov 14. PMID 29154779
- [Background] Zhuo Y, Cainuo S, Chen Y, Sun B. The efficacy of letrozole supplementation for medical abortion: a meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2021 May;34(9):1501-1507. doi: 10.1080/14767058.2019.1638899. Epub 2019 Jul 29. PMID 31257957
- [Background] Behroozi-Lak T, Derakhshan-Aydenloo S, Broomand F. Evaluation of effect of letrozole prior to misoprostol in comparison with misoprostol alone in success rate of induced abortion. J Gynecol Obstet Hum Reprod. 2018 Mar;47(3):113-117. doi: 10.1016/j.jogoh.2017.11.002. Epub 2017 Nov 6. PMID 29122709
- [Background] Naghshineh E, Allame Z, Farhat F. The effectiveness of using misoprostol with and without letrozole for successful medical abortion: A randomized placebo-controlled clinical trial. J Res Med Sci. 2015 Jun;20(6):585-9. doi: 10.4103/1735-1995.165964. PMID 26600834
- [Background] Rezai Z, Heydari Bazardehi S S, Ghasemi Nezhad A, Sadeghi A S, Ghorbani Yekta B. (2014). Letrozole and misoprostol versus misoprostol alone for termination of pregnancy: a randomized clinical trial. Tehran Univ Med J, 71 (11), 700-706
- [Background] Chawdhary R, Rana A, Pradhan N. Mifepristone plus vaginal misoprostol vs vaginal misoprostol alone for medical abortion in gestation 63 days or less in Nepalese women: a quasi-randomized controlled trial. J Obstet Gynaecol Res. 2009 Feb;35(1):78-85. doi: 10.1111/j.1447-0756.2008.00864.x. PMID 19215552
- [Background] Jain JK, Dutton C, Harwood B, Meckstroth KR, Mishell DR Jr. A prospective randomized, double-blinded, placebo-controlled trial comparing mifepristone and vaginal misoprostol to vaginal misoprostol alone for elective termination of early pregnancy. Hum Reprod. 2002 Jun;17(6):1477-82. doi: 10.1093/humrep/17.6.1477. PMID 12042265
- [Background] Blum J, Raghavan S, Dabash R, Ngoc Nt, Chelli H, Hajri S, Conkling K, Winikoff B. Comparison of misoprostol-only and combined mifepristone-misoprostol regimens for home-based early medical abortion in Tunisia and Vietnam. Int J Gynaecol Obstet. 2012 Aug;118(2):166-71. doi: 10.1016/j.ijgo.2012.03.039. Epub 2012 Jun 8. PMID 22682768
- [Background] Dahiya K, Ahuja K, Dhingra A, Duhan N, Nanda S. Efficacy and safety of mifepristone and buccal misoprostol versus buccal misoprostol alone for medical abortion. Arch Gynecol Obstet. 2012 Apr;285(4):1055-8. doi: 10.1007/s00404-011-2110-8. Epub 2011 Oct 19. PMID 22009509
- [Background] Fekih M, Fathallah K, Ben Regaya L, Bouguizane S, Chaieb A, Bibi M, Khairi H. Sublingual misoprostol for first trimester termination of pregnancy. Int J Gynaecol Obstet. 2010 Apr;109(1):67-70. doi: 10.1016/j.ijgo.2009.11.008. Epub 2010 Jan 6. PMID 20053398
- [Background] Ngoc NT, Blum J, Raghavan S, Nga NT, Dabash R, Diop A, Winikoff B. Comparing two early medical abortion regimens: mifepristone+misoprostol vs. misoprostol alone. Contraception. 2011 May;83(5):410-7. doi: 10.1016/j.contraception.2010.09.002. Epub 2010 Oct 18. PMID 21477682
- [Background] Allen R, O'Brien BM. Uses of misoprostol in obstetrics and gynecology. Rev Obstet Gynecol. 2009 Summer;2(3):159-68. PMID 19826573
- [Background] Chai J, Ho PC. A pilot study on the combined use of letrozole, mifepristone and misoprostol in termination of first trimester pregnancy up to 9 weeks' gestation. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):291-4. doi: 10.1016/j.ejogrb.2013.09.017. Epub 2013 Sep 25. PMID 24135383
- [Background] Yeung TW, Lee VC, Ng EH, Ho PC. A pilot study on the use of a 7-day course of letrozole followed by misoprostol for the termination of early pregnancy up to 63 days. Contraception. 2012 Dec;86(6):763-9. doi: 10.1016/j.contraception.2012.05.009. Epub 2012 Jun 18. PMID 22717187
- [Background] (Power Analysis and Sample Size Software (2015). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.)
- [Background] Lee VC, Tang OS, Ng EH, Yeung WS, Ho PC. A pilot study on the use of letrozole with either misoprostol or mifepristone for termination of pregnancy up to 63 days. Contraception. 2011 Jan;83(1):62-7. doi: 10.1016/j.contraception.2010.05.014. Epub 2010 Jun 23. PMID 21134505